CLINICAL TRIAL: NCT04496518
Title: Personalized Therapy Study - Intrinsic Antitachycardia Pacing Post-Approval Study (iATP PAS)
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: iATP PAS
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with ICD/CRT device with iATP programmed on: Patients implanted with an iATP-capable device with iATP on in at least one device detection zone will be enrolled in the iATP PAS. Patients must also be enrolled in the CareLink network for remote monitoring. All patients must have provided signed informed consent.
  Interventions: Device: Intrinsic Antitachycardia Pacing (iATP) Therapy

INTERVENTIONS:
Device: Intrinsic Antitachycardia Pacing (iATP) Therapy — iATP is a fully automated ATP therapy for monomorphic ventricular tachycardia (MVT).

SUMMARY:
Medtronic is sponsoring the Intrinsic Antitachycardia Pacing Post-Approval Study (iATP PAS) to further confirm safety and effectiveness of ventricular iATP therapy in routine clinical practice, following commercial release of iATP-capable devices.

The iATP PAS is conducted within Medtronic's Product Surveillance Registry platform (NCT01524276).

DETAILED DESCRIPTION:
The iATP PAS is a global, prospective, observational, multi-site registry study. Patients enrolled in the iATP PAS will be prospectively followed in the registry until registry closure, patient death, or patient exit from the registry (i.e., withdrawal of consent).

Patient and device status will be assessed at least annually or as prompted by reportable adverse events. Remote device data transmissions are recommended to occur at least quarterly. Primary objective analysis will occur when 241 iATP-treated eligible ventricular episodes in the fast ventricular tachycardia (FVT) zone have been collected and reviewed by the study episode review committee (ERC). The total study duration is approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient is intended to receive or is implanted with an iATP-capable device with iATP on in any zone with ventricular ATP therapies programmed.
* Patient is enrolled in the CareLink network for remote device monitoring

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients providing informed consent to participate prior to or within 30 days of implant of an iATP-capable cardiac rhythm device with iATP on in at least one zone. Patients need to be enrolled in Medtronic's CareLink network for remote device monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the success rate of iATP in the fast VT (FVT) zone is greater than 60% | Approximately 5 years
  Demonstrating success rate of iATP

SECONDARY OUTCOMES:
To demonstrate the success rate of iATP in the FVT zone is greater than 70% | Approximately 5 years
  Demonstrating success rate of iATP
To characterize arrhythmia-related syncope events | Approximately 5 years
  characterizing arrhythmia-related syncope events
To characterize unnecessary and inappropriate shocks | Approximately 5 years
  characterizing unnecessary and inappropriate shocks

CONTACTS AND LOCATIONS:
Locations (92):
- United States (51):
  - Southwest EP, Chandler, Arizona
  - Saint Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - Chula Vista Cardiac Center, Chula Vista, California
  - Cardiovascular Consultants Medical Group (Van Nuys CA), Van Nuys, California
  - Cardiology Associates Medical Group, Ventura, California
  - Colorado Springs Cardiology, Colorado Springs, Colorado
  - Denver Heart, Denver, Colorado
  - Colorado Heart and Vascular, PC, Lakewood, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Heart Rhythm Solutions, Hollywood, Florida
  - Baptist Health, Jacksonville, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Heart & Vascular Institute of Florida, Safety Harbor, Florida
  - Heart Rhythm Consultants P.A. (Sarasota Memorial Research), Sarasota, Florida
  - Deaconess Specialty Physicians, Evansville, Indiana
  - Iowa Heart Center (West Des Moines IA), Des Moines, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Norton Heart and Vascular Institute, Louisville, Kentucky
  - Tidal Health Peninsula Regional, Salisbury, Maryland
  - Associates in Cardiology PA, Silver Spring, Maryland
  - Brigham and Women's Hospital (Boston MA), Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Mayo Clinic (Rochester MN), Rochester, Minnesota
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - University Hospital (Columbia MO), Columbia, Missouri
  - Saint Lukes Health System, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Medicine, Omaha, Nebraska
  - Monmouth Cardiology Associates, Ocean City, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - South Shore University Hospital, Bay Shore, New York
  - Huntington Hospital, Huntington, New York
  - North Shore University Hospital, Manhasset, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - NewYork-Presbyterian/Columbia University Irving Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Staten Island University Hospital, Staten Island, New York
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - Summa Center for Clinical Trials-Northeast Ohio Cardiovascular Specialists, Akron, Ohio
  - The Christ Hospital Health Network, Cincinati, Ohio
  - St Luke's University Health Network, Bethlehem, Pennsylvania
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Heart Center of North Texas, Fort Worth, Texas
  - Consultants in Cardiology (Fort Worth TX), Fort Worth, Texas
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- France (11):
  - Clinique Rhône Durance, Avignon
  - CHU de Brest, Brest
  - Générale de Santé - Hôpital Privé Saint Martin, Caen
  - CHU de Caen - Hôpital Côte de Nacre - Centre Esquirol, Caen
  - CHU Clermont-Ferrand - Gabriel-Montpied, Clermont-Ferrand
  - CHU de Dijon - Hospital Le Bocage, Dijon
  - CHRU La Rochelle, La Rochelle
  - Nouvelles Cliniques Nantaises, Nantes
  - Centre hospitalier de la région d'Annecy, Pringy
  - Centre Hospitalier Universitaire Saint Étienne, Saint-Priest-en-Jarez
  - Capio - Clinique du Tonkin, Villeurbanne
- Greece (2):
  - Hygeia Hospital, Athens
  - Athens Medical Center, Marousi
- Italy (6):
  - Policlinico Sant' Orsola - Malpighi, Bologna
  - Azienda Sanitaria Provinciale di Cosenza"Ospedale di Castrovillari", Castrovillari
  - Ospedale "Vito Fazzi" Lecce, Lecce
  - Azienda Ospedaliera ospedale Niguarada ca Granda, Milan
  - Presidio Ospedaliero Centrale - SS.Annunziata, Taranto
  - Azienda ospedaleria Santa Maria dellaMisericordia di Udine, Udine
- Portugal (4):
  - Hospital da Senhora da Oliveira -Guimarães, Guimarães
  - Hospital de Santa Maria-Centro HospitalarLisboa Norte, EPE, Lisbon
  - Centro Hospitalar Universitário de SãoJoão Alameda, Porto
  - Hospital Distrital de Santarém, Santarém
- Národný ústav srdcových a cievnych chorôb, a.s. (NUSCH, a.s.), Bratislava, Slovakia
- Spain (8):
  - Hospital Universitario da coruna, A Coruña
  - Hospital Universitario Virgen de las Nieves, Granda
  - Hospital Universitario Clínico San Cecilio, Granda
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Universitario de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Switzerland (2):
  - Hôpitaux Universitaires de Genève, Geneva
  - Cardiopark Zurich, Zurich
- United Kingdom (7):
  - University Hospitals of Birmingham NHS Foundation Trust - Queen Elizabeth Hospital, Birmingham
  - Blackpool, Fylde and Wyre Hospitals NHSFoundation Trust - Blackpool Victoria Hospital, Blackpool
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Imperial College Healthcare NHS Trust Hammersmith Hospital, London
  - Central Manchester University Hospitals NHS - mancester Royal Infirmary, Manchester
  - The James Cook University Hospital - SouthTees Hospitals NHS, Middlesbrough
  - Sheffield Vascular Institute, Sheffield TeachingHospitals NHS - Northern Genera, Sheffield

IPD SHARING:
Plan to Share IPD: No